CLINICAL TRIAL: NCT06713902
Title: Fibrin Gel Loaded with Extracellular Vesicles for the Treatment of Cartilage Lesions in the Joints - GelVex Study
Brief Title: Extracellular Vesicles in Fibrin Gel for Cartilage Repair
Acronym: GelVex
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: GelVex
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Joint Disease
Keywords: Cartilage; Mesenchymal Stromal Cells; Extracellular Vesicles; Platelet Rich Plasma
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Fifty-one m/f patients matching the inclusion and exclusion criteria: Six patients undergoing plastic surgery procedures for the removal of adipose tissue from which waste material (adipose tissue) will be taken to obtain MSCs for EVs production. Five patients undergoing hip or knee joint replacement surgery from which waste material (osteo-cartilaginous material) will be taken to obtain chondrocytes for functional tests. Forty patients undergoing regenerative medicine treatments with PRP from which a waste aliquot (obtained during PRP preparation) will be taken to obtain plasma for fibrin gel production.

SUMMARY:
This project aims to produce and study in vitro/ex vivo a platelet rich plasma (PRP)-derived fibrin gel loaded with mesenchymal stromal cells (MSC)-extracellular vesicles (EVs), to combine the positive results on cartilage growth of PRP growth factors and the hyaline cartilage stimulating activity of MSC-EVs. Therefore, the project goal is to provide an advanced option for orthopedic patients with an innovative evolution of a gold standard procedure, making it easy to translate into daily clinical practice for physicians, healthcare professionals and patients.

ELIGIBILITY:
Inclusion Criteria:

* males and females ≥ 18
* patients undergoing plastic surgery procedures;
* patients undergoing elective joint surgery with a diagnosis of knee or hip osteoarthritis (any Kellgren-Lawrence grade);
* patients undergoing regenerative medicine treatments with PRP with a diagnosis of knee or hip osteoarthritis (any Kellgren-Lawrence grade;
* signed Informed Consent for the study

Exclusion Criteria:

* Positive virological test (HIV, HCV, HBV, TPHA)
* Pregnancy or breastfeeding by self-declaration
* Other conditions that, at the discretion of the investigator or the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Upon signing the Informed Consent, 51 male and female subjects, ≥ 18 years old, attending the IRCCS Galeazzi-Sant'Ambrogio Hospital and matching the inclusion and esclusion criteria will be recruited.
Sampling Method: Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Confirm the incorporation rate of extracellular vesicles (EV) into platelet-rich plasma (PRP) following the formation of fibrin gel | 2 years
  To implement the preliminary data obtained by the PI in the development of a protocol to achieve efficient incorporation of mesenchymal stem cell-derived extracellular vesicles into platelet-rich plasma-derived fibrin gels and characterize their release. MSC-EVs will be embedded in fibrin gel using PRP provided by patients enrolled in the study that is activated to obtain the solid form. To monitor the incorporation and release of EVs from the PRP-gel, EVs will be labeled with a fluorescent marker to allow their subsequent detection by cytometry or imaging methods. The ability of the released EVs to be incorporated into human chondrocytes and penetrate cartilage will be tested using three in vitro models: i) flow cytometry in a 2D culture model; ii) a 3D microfluidic model; iii) a Quantitative Imaging with cartilage explants. Biological activity will be tested on pathological chondrocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ragni E, De Luca P, Landoni S, Valli F, Mortati L, Palombella S, Talo G, Moretti M, de Girolamo L. High efficiency protocol for platelet derived fibrin gel loaded with mesenchymal stromal cells extracellular vesicles. Regen Ther. 2024 Jul 7;26:442-457. doi: 10.1016/j.reth.2024.06.020. eCollection 2024 Jun. PMID 39070124